CLINICAL TRIAL: NCT05121428
Title: Exploring the Attitudes and Experiences of Patients Engaged in Buprenorphine Treatment During the COVID-19 Pandemic
Brief Title: Patients' Attitudes Toward and Experiences With Buprenorphine Treatment
Status: Suspended | Type: Observational
Why Stopped: Study completed Phase 1 before funding ended.
Sponsor: Cambridge Health Alliance (Other)
Collaborators: National Cancer Institute (NCI) (NIH); National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Other Study IDs: CHA-IRB-1179/03/21; 3R33AT010125 (NIH); R01CA229355 (NIH)
Record Dates: First submitted 2021-10-21; First posted 2021-11-16 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-06

CONDITIONS: Opioid-use Disorder; Acceptability of Health Care; Opioid-Related Disorders
Keywords: Opioid Use Disorder; Substance Use Disorders; Buprenorphine; Suboxone; Cannabis; Cigarettes; E-Cigarettes; Benzodiazepines; Healthcare; COVID-19; Telemedicine; Office-Based Opioid Treatment; Facebook; Social Media; Nicotine; Recovery
MeSH Terms: conditions — Opioid-Related Disorders; Patient Acceptance of Health Care; Substance-Related Disorders; Marijuana Abuse; Vaping; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (5):
- Survey 1: Survey investigating patients' experiences with buprenorphine treatment for Opioid Use Disorder before and during the COVID-19 pandemic
- Survey 2: Survey investigating the factors that motivate patients to abstain from opioid drug use during buprenorphine treatment for Opioid Use Disorder
- Survey 3: Survey investigating patients' attitudes towards and experiences with cannabis use during buprenorphine treatment for Opioid Use Disorder.
- Survey 4: Survey investigating patients' attitudes towards and experiences with cigarettes and e-cigarettes use during buprenorphine treatment for Opioid Use Disorder.
- Survey 5: Survey investigating patients' attitudes towards and experiences with benzodiazepine use during buprenorphine treatment for Opioid Use Disorder.

SUMMARY:
This study will disseminate five surveys collecting individual's attitudes and experiences during buprenorphine treatment for Opioid Use Disorder during the COVID-19 pandemic.

DETAILED DESCRIPTION:
The primary objective of this study is to better understand patients' attitudes and experiences during office-based opioid treatment (OBOT) in the COVID-19 pandemic. This study specifically aims to evaluate attitudes and experiences of people prescribe buprenorphine across five domains with the hope of evaluating a) whether telemedicine has improved their access to and experiences with OBOT; b) the factors that motivate individuals in OBOT to abstain from opioid drug use; c) how patients' view the use of cannabis, benzodiazepines, and nicotine during OBOT; d) the degree to which patients in OBOT report using cannabis, benzodiazepines, and nicotine and how their use might have changed during the COVID-19 pandemic; and e) whether patients attitudes towards cannabis, benzodiazepines, and cigarettes/e-cigarettes are associated with their use of those same substances.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be 18 years of age or older.
* Participants report currently having a legal prescription for buprenorphine for opioid use disorder.
* Participants must have a past or present opioid use disorder.
* Participants must currently reside in the state of Massachusetts.
* Participants must be able to comprehend the English language.

Exclusion Criteria:

* Unable to complete an online survey.
* Unable to complete a verification step that ensures bots are not used to complete survey.
* Complete a survey with no variation suggesting they did not read the survey.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The subject population consists of adults aged 18+ who live in Massachusetts and are currently prescribed buprenorphine by a healthcare provider to treat OUD. Those under the age of 18 will be screened out of the investigation during the consent process. In addition, because many of the survey questions used in this investigation are based on established survey instruments that were created in the English language and validated among English-speaking participants, we will limit the subject population or this study to English-speaking adults.
Sampling Method: Non-Probability Sample
Enrollment: 817 (Actual)
Dates: Start 2021-11-20 (Actual); Primary Completion 2025-03-20 (Actual); Study Completion 2027-03-20 (Estimated)

PRIMARY OUTCOMES:
Patient's Experiences with Office-Based Opioid Treatment | Day 1
  This is an eight-item scale that measures the degree to which participants report being able to access buprenorphine treatment-related appointments and medications before and during the COVID-19 pandemic. Participants will be asked to rate each of the eight questions on a 7-point Likert scale from 1 = "extremely easy" to 7= "extremely difficult."
Reasons for Abstaining from Opioids Questionnaire | Day 1
  This 17-item scale will measure participant ratings of the importance of 17 factors that motivate abstinence from illicit drug use during office-based opioid treatment. Participants will be asked to rate each of these 17 items on a scale from 0 = "not at all important" to 4 = "extremely important."
Patients' Attitudes Toward the Use of Cannabis During Office-Based Opioid Treatment | Day 1
  Participants will rate three items on a scale of 1 = "completely disagree" to 7 = "completely agree." Specifically, participants will rate the degree to which they feel cannabis use is acceptable during office-based opioid treatment (OBOT), they believe that their prescribers' feel cannabis use is acceptable during OBOT, and they feel comfortable discussing cannabis use with their buprenorphine prescribers.
Patients' Attitudes Toward the Use of Cigarettes/E-Cigarettes During Office-Based Opioid Treatment | Day 1
  Participants will rate three items on a scale of 1 = "completely disagree" to 7 = "completely agree." Specifically, participants will rate the degree to which patients should be encouraged to quit smoking cigarettes and e-cigarette during office-based opioid treatment (OBOT) and the degree to which they feel smoking helps manage cravings during OBOT.
Patients' Attitudes Toward and Experiences with the Use of Benzodiazepines during Office-Based Opioid Treatment | Day 1
  Participants will rate three items on a scale of 1 = "completely disagree" to 7 = "completely agree." Specifically, participants will rate the degree to which benzodiazepine use is acceptable during office-based opioid treatment (OBOT), they feel OBOT providers find benzodiazepine use by their patients acceptable, and they feel comfortable openly discussing their benzodiazepine use with their buprenorphine prescriber.

CONTACTS AND LOCATIONS:
Overall Officials: Zev Schuman-Olivier, MD, Principal Investigator — Cambridge Health Alliance; Joseph Rosansky, Study Director — Cambridge Health Alliance
Locations (1):
- CHA Center for Mindfulness and Compassion, Cambridge, Massachusetts, United States